CLINICAL TRIAL: NCT02232295
Title: To Study the Effect of Graded Motor Imagery on Upper Limb Motor Functions and Quality of Life in Patients With Stroke
Brief Title: A Clinical Trial to Study the Effect of Imagined Progressive Movements in Patients With Paralysis of One Side of the Body.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Manisha Uttam, Physiotherapist, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M44-124
Record Dates: First submitted 2014-08-29; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Stroke
Keywords: Upper extremity, motor imagery, mirror therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional group (Active Comparator): Conventional group consist of Upper extremity task oriented functional exercises. Components of Task oriented training include weight bearing, supportive reactions, and reaching, grasping, holding and release activities.
  Interventions: Device: Mirror Box
- Graded Motor imagery group and Conventional group (Experimental): Graded Motor imagery is a three stage process, was performed five days a week for six weeks of one hour duration. It comprises of:
  * Left Right discrimination training (Implicit Motor Imagery) - 2 weeks
  * Explicit Motor Imagery (Imagined movements) - 2 weeks
  * Mirror Therapy - 2 weeks
  Interventions: Device: Recognise [TM]

INTERVENTIONS:
Device: Recognise [TM] — Recognise accurately measures to identify left and right body parts and movements, and to train left/right discrimination as part of a comprehensive GMI rehabilitation process.
  Other Names: Online Recognise software by the NOI group, Australia
  Arms: Graded Motor imagery group and Conventional group
Device: Mirror Box — A resource used for many pain and disability states of the hands and feet.
  Arms: Conventional group

SUMMARY:
The aim of the Study to evaluate the effect of Graded motor imagery on upper limb motor functions and quality of life in patients with stroke that was conducted in two centers in india. The primary outcome measures were upper limb motor functions at 6 weeks and secondary outcome measure was quality of life at 6 weeks.

Research Hypothesis: There would be significant effect of GMI on Upper limb motor functions and quality of life in patients with stroke.

DETAILED DESCRIPTION:
Graded Motor Imagery (GMI) is essentially a brain based treatment, targeting the activation of different brain regions in a graded manner. GMI is a three stage treatment programme comprising of Left Right discrimination training, Explicit Motor imagery and Mirror therapy.

In this Study, GMI approach is applied on the patients with Stroke to enhance their Upper limb motor functions and Quality of life.

Conventional treatment:

Patients of group A and group B had received conventional treatment for 6 weeks. Conventional treatment consists of Task oriented upper extremity functional exercises. Components of Task oriented training include weight bearing, supportive reactions, and reaching, grasping, holding and release activities. It was performed five days a week for six weeks of one hour duration.

Graded Motor Imagery:

Patients of group A had received GMI programme with conventional treatment for 6 weeks. It is a three stage process, was performed five days a week for six weeks of one hour duration. It comprises of:

* Left Right discrimination training (Implicit Motor Imagery) - 2 weeks
* Explicit Motor Imagery (Imagined movements) - 2 weeks
* Mirror Therapy - 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age (between 45 to 65 years)
* Individuals who experienced one episode of stroke only.
* Both males and females were included in the study
* Both ischemic & haemorrhagic stroke individuals were included in the study
* Duration of stroke between 1 to 6 months
* Mini mental status examination (MMSE) (score > 23)
* Patients with Brunnstrom stage 1 & 2

Exclusion Criteria:

* Individuals having any musculoskeletal disorders
* Individuals having any neurological disorder other than stroke
* Individuals with any visual impairment
* Individuals having any systemic disease
* Non cooperative patients
* Patients suffering from psychological problems

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Upper limb motor functions | six weeks
  Primary Outcome measures: FMA Scale and CAHAI scale
  FMA Scale:
  It is a stroke specific, performance based impairment index. This scale includes items related to movements of the shoulder, elbow, forearm, wrist, and hand in the upper extremity, as well as the hip, knee, and ankle in the lower extremity. For the present study, only the upper extremity was measured.The total score on the upper extremity part of the FMA ranged from 0 (hemiplegia) to a maximum of 66 points (normal motor performance). The scale was measured at baseline and post intervention.
  CAHAI Scale:
  The purpose of this measure is to evaluate the functional ability of the hemiplegic arm and hand to perform tasks. It is designed to encourage the bilateral hand to complete the task.Each task was demonstrated once before performance, then the Score was evaluated of the affected upper extremity using the 7 point activity scale from total assistance (1) to complete

SECONDARY OUTCOMES:
Quality of life | 6 weeks
  Secondary outcome measure:
  SS-QOL (Stroke Specific- Quality of life) Scale It is a self report scale containing 49 items in 12 domains. It is intended to provide an assessment of health related quality of life specific to patients with stroke. Scale domains and items were derived from a series of interviews with patients.The scale was measured at baseline and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Uttam, Masters in Physiotherapy, Principal Investigator — Maharishi Markandeshwar University, Mullana-Ambala
Locations (1):
- Maharishi Markandeshwar institute of Physiotherapy and rehabilitation, MMU, Mullana, Ambāla, Haryana, India